CLINICAL TRIAL: NCT07116473
Title: A Phase 3, Open-Label, Multicenter, Extension Study of Acoramidis in Patients With Newly Diagnosed Variant Transthyretin Amyloid Cardiomyopathy (ACT-EARLY OLE)
Brief Title: To Evaluate the Long-term Safety and Tolerability of Acoramidis in Participants With Newly Diagnosed ATTR-CM (ACT-EARLY OLE)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eidos Therapeutics, a BridgeBio company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AG10-504; U1111-1323-6219 (WHO) (Other: WHO); 2024-513676-18-00 (EUCT) (Other: EUCT)
Record Dates: First submitted 2025-08-07; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Amyloidosis in Transthyretin (TTR); Amyloidosis, Familial; Amyloid Cardiomyopathy; Amyloid Cardiomyopathy, Transthyretin-Related; Amyloidogenic Transthyretin (ATTR) Amyloidosis; Heart Disease; Cardiomyopathies; Amyloidosis, Hereditary, Transthyretin-Related; Polyneuropathies; Amyloidosis
Keywords: ATTR-CM; ATTR-PN; Amyloidosis; Transthyretin; Amyloid; TTR; Hereditary
MeSH Terms: conditions — Amyloidosis, Familial; Amyloid Neuropathies, Familial; Amyloidosis; Heart Diseases; Cardiomyopathies; Amyloidosis, Hereditary, Transthyretin-Related; Polyneuropathies; Alzheimer Disease | interventions — attruby

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Acoramidis (Experimental): Participants will receive acoramidis 712 mg orally BID (which is equivalent to 800 mg acoramidis HCl BID)
  Interventions: Drug: Acoramidis (AG10)

INTERVENTIONS:
Drug: Acoramidis (AG10) — TTR stabilizer administered orally twice daily (BID)
  Other Names: ALXN2060

SUMMARY:
The AG10-504 study is an open-label extension study of acoramidis in participants with newly diagnosed transthyretin amyloid cardiomyopathy (ATTR-CM) or both ATTR-CM and transthyretin amyloid polyneuropathy (ATTR-PN).

DETAILED DESCRIPTION:
The AG10-504 study is the extension of the Phase 3 AG10-501 study (ACT-EARLY) which was designed to investigate if the use of acoramidis as a prophylactic intervention in individuals who are carriers of a known pathogenic transthyretin (TTR) variant but with no clinical evidence of ATTR could prevent or delay the onset of clinically detectable ATTR and the considerable morbidity and mortality that result from this devastating, progressive, and ultimately fatal disease. Only participants who have completed the AG10-501 study (ACT-EARLY) with a diagnosis of ATTR-CM may enroll in this AG10-504 Open Label Extension (OLE) study.

The primary objective of the AG10-504 study is to evaluate the long-term safety and tolerability of acoramidis in participants with newly diagnosed ATTR-CM. The duration of this study will be up to 5 years.

Currently, acoramidis is approved for the treatment of ATTR-CM in some regions including the United States, United Kingdom, Japan, and the European Union.

ELIGIBILITY:
Key Inclusion Criteria:

Participants must have completed the AG10-501 study (ACT-EARLY study) within the past 60 calendar days with a diagnosis of ATTR-CM (based on the AG10-501 protocol definition of ATTR-CM).

Key Exclusion Criteria:

1. Participants who completed the AG10-501 study with a diagnosis of ATTR-PN only, or who permanently discontinued study drug prior to diagnosis of ATTR-CM in AG10-501.
2. History of AL or another non-TTR amyloid subtype (eg, ApoA-1, gelsolin).
3. History of a monoclonal paraprotein or abnormal light chains in serum or urine (i.e., MGUS) in which AL has not been ruled out.
4. Stage IV or V chronic kidney disease (corresponding to an eGFR ≤ 29 mL/min/1.73 m2), or undergoing renal dialysis, or recipient of a kidney transplant.
5. Active malignancy, except for basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix that has been successfully treated. In the event a participant developed a low-grade and treatable malignancy in the AG10-501 study (eg, low-grade, localized prostate cancer) and the decision by the Investigator at that time was to continue the participant in the AG10-501 study, that participant may still qualify for Study AG10-504 after documentation with the Medical Monitor.
6. History of any organ transplant (with the exception of corneal transplant).
7. Known hypersensitivity to acoramidis or any of the excipients within the study drug.
8. Treatment for ATTR-CM with any ATTR-oriented on- or off-label or OTC product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2037-11 (Estimated); Study Completion 2037-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the long-term safety and tolerability of acoramidis in participants with newly diagnosed ATTR-CM | The duration of study participation for the participants will be up to 5 years.
  Proportion of participants with: treatment-emergent AEs and SAEs, AEs leading to treatment discontinuation, abnormal physical examination findings of clinical relevance, abnormal vital signs of clinical relevance, abnormal ECG parameters of clinical relevance, changes in clinical safety laboratory parameters of potential concern